CLINICAL TRIAL: NCT01240343
Title: Creation of the Biobank Related to Eye Disease
Acronym: BioBank
Status: Completed | Type: Observational
Sponsor: Kimberly Drenser (Other)
Collaborators: Vision Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Kimberly Drenser, M.D, Ph.D., Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2009-057
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Eye Diseases
Keywords: Biobank; Genetics
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine other body fluids (i.e. vitreous)
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a BioBank (a specialized lab) and collect blood, fluids and/or other tissue samples to study eye diseases.

DETAILED DESCRIPTION:
The purpose of the Biobank related to eye disease at Beaumont Hospital is to help connect specialties and Specialists with each other, outside traditional limits of hospital or laboratory departments. The specimens (blood, fluids, and/or tissue samples) that will be collected from men, women and children will assist the researchers in a variety of studies on human eye diseases.

Research utilizing these specimens will allow for an increased understanding of the etiology, disease process, and response to treatments for various eye diseases, and will provide opportunities to subsequently improve our management decisions. Furthermore, projects that cross over between subspecialties are sparse and that is a limiting factor for the development of research that takes a more comprehensive approach.

ELIGIBILITY:
Inclusion Criteria: All pediatric and adult patients age 0-99 years -

Exclusion Criteria: All patients who do not agree to consent for collection of blood, fluids, tissue.

Patients who are cognitively impaired and are not able to verbalize understanding of the risks/benefits.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pediatric and adult patients (age 0-99)who are being seen in the eye Dr. office and or having eye surgery
Sampling Method: Non-Probability Sample
Enrollment: 669 (Actual)
Dates: Start 2009-06; Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
To build the platform for a novel application of translational research that links cutting edge molecular laboratory techniques to clinical outcome studies
  Biobanks can be used for numberous discovery applications such as: identification and structural characterization of human genes, expression analysis, or discovery proteomics. Biological specimens, when coupled with standardized treatment and outcome data, will be essential resources for the identification, characterization and validation of biomarkers that are predictive of disease and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Drenser, MD, PhD, Principal Investigator — Associated Retinal Consultants, P.C.
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share at this time